CLINICAL TRIAL: NCT00795509
Title: Special Investigation For Long Term Use Of Detrusitol (Regulatory Post Marketing Commitment Plan).
Brief Title: Special Investigation For Long Term Use Of Tolterodine (Regulatory Post Marketing Commitment Plan).
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6121187
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-06

CONDITIONS: Urinary Bladder, Overactive
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tolterodine tartrate.: Patients taking Tolterodine tartrate.
  Interventions: Drug: Tolterodine tartrate

INTERVENTIONS:
Drug: Tolterodine tartrate — Detrusitol® Capsule 2mg and 4mg, depending on the Investigator prescription. Frequency and duration are according to Package Insert as follows. " The usual adult dosage for oral administration is 4 mg of tolterodine tartrate once daily. Occasionally dose reduction might be needed due to individual tolerability."
  Other Names: Detrusitol® Capsule.

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the LPD (unknown adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3)factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Detrusitol® Capsule should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be administered Detrusitol® Capsule in order to be enrolled in the surveillance.

Exclusion Criteria:

* Patients not administered Detrusitol® Capsule.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A6121187 prescribes the Tolterodine tartrate (Detrusitol® Capsule).
Sampling Method: Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2007-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6121187&StudyName=Special%20Investigation%20For%20Long%20Term%20Use%20Of%20Tolterodine%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29.

RESULTS

PARTICIPANT FLOW:
Groups:
- Tolterodine Tartrate.: Participants taking Tolterodine tartrate.
Period: Overall Study
Arm/Group | Tolterodine Tartrate.
Started | 374
Completed | 343
Not Completed | 31
Not completed — Protocol Violation | 31

BASELINE CHARACTERISTICS:
Arm/Group | Tolterodine Tartrate.
Number analyzed (Participants) | 343
Age, Customized [Number; unit: participants]
  <65 years | 98
  >= 65 years | 245
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159
  Male | 184
Target disease severity [Number; unit: participants] — The severity of Overactive Bladder which was diagnosed by investigator.
  participants
    Mild | 135
    Moderate | 194
    Severe | 14
Complications [Number; unit: participants]
  Present | 266
  Absent | 77
Concomitant drug [Number; unit: participants]
  Present | 256
  Absent | 87
Treatment Period [Number; unit: participants]
  Less than 12 weeks | 1
  12 to 24 weeks | 44
  24 to 52 weeks | 88
  52 to 76 weeks | 172
  76 to 104 weeks | 31
  Over 104 weeks | 7

OUTCOME MEASURES:

1. Primary Outcome: Adverse Drug Reaction Not Expected From the Japanese Package Insert. Number of Unlisted Treatment Related Adverse Events (TRAEs).
Description: All observed or volunteered adverse events and the investigator's opinion of the causal relationship to the study treatment were reported. Definition of an adverse event (AE) is any adverse change in health or side effect that occurs in participates. Treatment related Adverse Events were evaluated in company with the causal relationship to the investigational product. Unlisted treatment related adverse events were confirmed with listed adverse drug reaction in Japanese package insert.
Time Frame: 52 weeks
Population: Safety analysis population included all enrolled participants who had received at least 1 confirmed, administration of Detorsitol.
Measure: Number; unit: participants
Arm/Group | Tolterodine Tartrate.
Number analyzed (Participants) | 343
participants
  Glaucoma | 1
  Death | 1
  Abdominal discomfort | 1

2. Primary Outcome: Confirmation of the Incidence of All Treatment Related Adverse Events (TRAEs).
Description: All observed or volunteered adverse events and the investigator's opinion of the causal relationship to the study treatment were reported. Definition of an adverse event (AE) is any adverse change in health or side effect that occurs in participates. Treatment related Adverse Events were evaluated in company with the causal relationship to the investigational product.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Tolterodine Tartrate.
Number analyzed (Participants) | 343
participants | 25

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tolterodine Tartrate.
Serious Adverse Events (participants affected / at risk) | 1/343
Other Adverse Events (participants affected / at risk) | 25/343
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolterodine Tartrate. (N=343)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolterodine Tartrate. (N=343)
Dysuria (Renal and urinary disorders) | 8 (8)
Constipation (Gastrointestinal disorders) | 6 (6)
Thirst (General disorders) | 6 (6)
Urinary retention (Renal and urinary disorders) | 4 (4)
Residual urine volume increased (Renal and urinary disorders) | 3 (3)
Dizzines (Nervous system disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.